CLINICAL TRIAL: NCT07058909
Title: Premarket Clinical Safety Assessment of the ELISIO™-HX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nipro Medical Corporation (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMC-PRO-0009
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Renal Failure; Acute Renal Failure; Chronic Renal Failure; Chronic Kidney Diseases; End Stage Renal Disease
Keywords: Hemodialyzer; High-permeability hemodialyzer; Expanded hemodialysis (HDx); Expanded solute removal; Medium cutoff (MCO) dialyzer; Dialysis
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury; Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ELISIO™-HX Dialyzer (Experimental): The ELISIO™-HX is a single use novel medium cut-off dialyzer that is intended for use as an artificial kidney for the treatment of participants with renal failure.
  Interventions: Device: ELISIO™-HX Dialyzer

INTERVENTIONS:
Device: ELISIO™-HX Dialyzer — Following consent, participants will undergo a baseline hemodialysis treatment with their currently used dialyzer, the ELISIO-H™, and following the baseline visit will receive hemodialysis with the investigational device, ELISIO™-HX, three times a week for 12 weeks.

SUMMARY:
The primary safety objective of this study is to evaluate the safety of the use of the high-permeability hemodialyzer series ELISIO™-HX, by showing that the pre-dialysis albumin levels are not affected using the investigational dialyzer.

The primary efficacy objective is to evaluate the performance of the use of the high permeability hemodialyzer series ELISIO™-HX, by showing that the clearance rate of middle molecular weight lambda (λ) free light chain (FLC) is improved by using the investigational dialyzer.

ELIGIBILITY:
Inclusion Criteria:

1. End stage renal disease patients on hemodialysis age 22 and older, or between ages 18 and 21 with a weight ≥40 kg.
2. Clinically stable as judged by the treating physician and as demonstrated by stable medical history for 30 days prior to enrollment, physical examination, and laboratory testing.
3. Hemodialysis therapy with the ELISIO-H dialyzer for at least 3 months immediately prior to study enrollment and expected to survive for the next 12 months.
4. Expected to maintain an acceptable urea clearance (Kt/V) with a dialyzer of an approximate surface area of 1.7 m2.
5. Currently being dialyzed at an in-center setting, on a schedule of 3 times per week.
6. Able to give informed consent after an explanation of the proposed study, and willing to comply with the study requirements for therapy during the entire study treatment period.
7. Have a stable functioning vascular access (arteriovenous fistula, graft, or dual lumen tunneled catheter). Stable access should be confirmed by:

   1. Kt/V ≥1.2 for past 2 measurements, and/or
   2. Achievement of within 15% the prescribed blood flow rate (≥350 ml/min) over 3 treatments prior to study entry Note: must have a flow of ≥350 ml/min at the time of enrollment.
8. Participants who have given their informed consent in writing.

Exclusion Criteria:

1. Are female and pregnant, lactating, or planning to become pregnant during the study period. Note: Female participants of childbearing potential, defined as a woman <55 years old who has not had a partial or full hysterectomy or oophorectomy, must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test at screening. Participants of childbearing potential must use a medically acceptable means of contraception during their participation in the study.
2. Have chronic liver disease.
3. Have a known paraprotein-associated disease.
4. Have known bleeding disorders (e.g., gastrointestinal bleeding, colonic polyps, small bowel angiodysplasia, and active peptic ulcers).
5. Have had a major bleeding episode (e.g., soft tissue bleeding, blood in stool, prolonged nose bleeds, joint damage, retinal bleeding, extensive mucosal bleeding, exsanguination, cerebral hemorrhage) ≤12 weeks prior to enrolling.
6. Have had a blood (red blood cell) transfusion ≤12 weeks prior to enrollment.
7. Have had an acute infection ≤4 weeks prior to enrollment.
8. Have active cancer, except for basal cell or squamous cell skin cancer.
9. Have a known serum κ/λ FLC ratio that is less than 0.37, or greater than 3.1
10. Have a known monoclonal gammopathy (monoclonal gammopathy of uncertain significance, smoldering [asymptomatic] multiple myeloma, symptomatic multiple myeloma, plasmacytomas, or plasma cell leukemia).
11. Have a known polyclonal gammopathy (connective tissue disease, liver disease, chronic infection, lymphoproliferative disorder, or other hematologic condition).
12. Have a positive serology test for human immunodeficiency virus or hepatitis infection.
13. Have a significant psychiatric disorder or mental disability.
14. Are scheduled for planned interventions requiring hospitalization >1 week.
15. Are scheduled for living-donor transplantation within the study period + 3 months, plan to change to peritoneal dialysis (PD) therapy within the next 9 months, plan to change to a home hemodialysis treatment, or plan to relocate to an area where no study center is located.
16. Are currently participating in another interventional clinical study or have participated in another interventional clinical study in the past 3 months.
17. Have a history of non-compliance with HD as assessed by an investigator.
18. Have had a major cardiovascular or cerebrovascular event within 3 months of enrollment.
19. Have a history with consistent evidence of intradialytic hypotension.
20. Have uncontrolled (systolic BP > 180 mmHg) hypertension.
21. Have had adverse reactions to dialyzer materials
22. Vulnerable participant populations (e.g., incarcerated or cognitively challenged adults)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in serum level of albumin | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks of treatment with ELISIO-HX
Reduction ratio (RR) of lambda (λ) FLC | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks of treatment with ELISIO-HX

SECONDARY OUTCOMES:
Change in Factor VII | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks
Change in Protein C | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks
Change in Factor II | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks
Change in Vitamin A | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks
Change in nPNA(nPCR) [normalized Protein equivalent of Nitrogen Appearance (normalized Protein Catabolic Rate)] | Baseline (last blood draw post-dialysis with ELISIO-H) to last blood draw post-dialysis after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiranjit Dhillon, MD, MPH, Principal Investigator — Davita Norfolk Dialysis Center
Locations (1):
- Davita Clinical Research, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No